CLINICAL TRIAL: NCT03204513
Title: Impact of Powered Knee-Ankle Prosthesis Leg on Everyday Community Mobility and Social Interaction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Arun Jayaraman, PT, PhD, Principal Investigator, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00200842
Record Dates: First submitted 2017-06-22; First posted 2017-07-02 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Transfemoral Amputees
Keywords: Prosthesis; Powered Prosthesis
MeSH Terms: interventions — Knee Prosthesis

STUDY DESIGN:
Intervention Model Description: Upon screening and enrollment participants return for up to 8 prosthetic fitting sessions and up to 12 physical therapy training sessions using their own microprocessor (MP) knee prosthesis and the powered knee-ankle (PKA) prosthesis. Once training is complete participants will return for up to 6 post-training assessment sessions per device. The device participants begin with will be randomly selected but there will be equal opportunity to train with both devices. In between training, there will be an 8 week "wash out period" to allow normalization to use of the device, reducing carryover effects. After wash-out period protocol will be repeated with second device.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vanderbilt Powered Knee-Ankle Prosthesis (Experimental): Upon screening and enrollment participants return for up to 8 prosthetic fitting sessions and up to 12 physical therapy training sessions using the Vanderbilt Powered Knee-Ankle (PKA) Prosthesis. Once training is complete participants will return for up to 6 post-training assessment sessions using the Vanderbilt Powered Knee-Ankle (PKA) Prosthesis. The device participants begin with will be randomly selected but there will be an equal opportunity to train with both devices. In between training, there will be an 8 week "wash out period" to allow normalization to use of the device, reducing carryover effects. After wash-out period protocol will be repeated with second device.
  Interventions: Device: Vanderbilt Powered Knee-Ankle Prosthesis
- Microprocessor (MP) Knee Prosthesis (Active Comparator): Upon screening and enrollment participants return for up to 8 prosthetic fitting sessions and up to 12 physical therapy training sessions using their own Microprocessor (MP) Knee Prosthesis. Once training is complete participants will return for up to 6 post-training assessment sessions using the Microprocessor (MP) Knee Prosthesis. The device participants begin with will be randomly selected but there will be an equal opportunity to train with both devices. In between training, there will be an 8 week "wash out period" to allow normalization to use of the device, reducing carryover effects. After wash-out period protocol will be repeated with second device.
  Interventions: Device: Microprocessor (MP) Knee Prosthesis

INTERVENTIONS:
Device: Vanderbilt Powered Knee-Ankle Prosthesis — The Vanderbilt powered prosthesis is a transfemoral prosthesis with powered and coordinated knee and ankle joints. The Generation 3 prosthesis is actuated by two brushless direct current (DC) motors, providing up to 100 Nm of torque at the knee joint, and with the assistance of a parallel stiffness, up to 200 Nm in plantar flexion at the ankle. Sensors measure knee and ankle joint angles, axial load in the shank, and position and orientation of the prosthesis in space (via a 6-axis inertial measurement unit). An onboard lithium-ion battery provides sufficient energy for approximately 10,000 steps between battery charges. The prosthesis prototype weighs approximately 4.3 kg (9.5 lb), the mass of which is approximately equivalent to the intact limb of a 48 kg (105 lb) person.
  Other Names: PKA Prosthesis; Powered Knee-Ankle Prosthesis
  Arms: Vanderbilt Powered Knee-Ankle Prosthesis
Device: Microprocessor (MP) Knee Prosthesis — Participants enrolled will already have their own microprocessor controlled (MP) non-powered knee prostheses as per inclusion criteria. Examples: OttoBock's C-Leg, Ossur's Rheo, Freedom Plie, Endolite Orion,etc.
  Arms: Microprocessor (MP) Knee Prosthesis

SUMMARY:
The overall goal of this research is to determine the efficacy of new powered prosthetic devices for individuals with transfemoral amputations. The anticipation is that this will be a high-impact technological intervention with the potential to restore significant functionality to individuals with lower limb amputation and transform the field of lower limb prosthetics. The objective of the proposed clinical trial is to fully evaluate the biomechanical and energetic effects of using PKA prosthesis and quantify functional performance and quality of life changes.

DETAILED DESCRIPTION:
The overall goal of this research is to bring powered devices, with suitable advanced control systems, to the clinic and home. The anticipation is that this will be a high-impact technological intervention with the potential to restore significant functionality to individuals with lower limb amputation and transform the field of lower limb prosthetics.

The objective of the proposed clinical trial is to fully evaluate the biomechanical and energetic effects of using a powered knee-ankle prosthesis, identify task-specific training strategies for every-day device use, and quantify functional performance and quality of life changes at home and in the community. The hypothesis is that the powered knee-ankle prosthesis will demonstrate a significant improvement in function over existing technology. Furthermore, the hypothesis is that incorporating neural control information will provide enhanced, intuitive control of this device. Thus the approach is to directly compare the powered device with current state-of-art passive microprocessor controlled (MP) prostheses using a randomized cross-over study to control for subject-specific variation.

1.1 Aim 1: Perform in-laboratory training and testing to compare gait biomechanics and clinical performance over several ambulation modes using either a passive prosthesis or a powered prosthesis. The expectation is the PKA prosthesis to enable gait kinetics and kinematics that more closely resemble those of individuals with intact limbs, therefore lowering the biomechanical and metabolic effects of ambulation.

1.2 Aim 2: Perform home trials to evaluate community mobility and social interaction when using a powered knee-ankle prosthesis or a passive device. The expectation is that participants will choose to complete more diverse functional, occupational, and recreational activities when using the PKA prosthesis.

1.3 Aim 3: Quantify performance with the PKA device when using a novel intent recognition algorithm that allows for seamless transitioning between activities compared to a standard control method. The expectation is that pattern recognition- based control will further improve mobility and decrease the physiological costs of ambulation compared to using the standard control method.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral level limb loss or limb difference
* K2/K3/K4 level ambulators
* Required to use a microprocessor knee on their prosthesis

Exclusion Criteria:

* Over 250 lbs body weight
* Inactive, physically unfit
* Cognitive deficits or visual impairment that would impair their ability to give informed consent or to follow simple instructions during the experiments
* Pregnant women
* Co-morbidity that interferes with the study (e.g. stroke, pace maker placement, severe ischemia cardiac disease, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change between devices of the Modified Graded Treadmill Test | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  This test is used to determine participant's endurance while walking at different speeds on a motorized treadmill. Participants will be secured to an overhead safety harness during this test. Participants will walk for up to 2 minutes each at different speeds on the treadmill. The treadmill speeds will be varied between 0.2 meters/second up to 2.0 meters/second at increments of 0.2 meters/sec. Close to the end of every 2 minute walk period, the participant will be asked to rate the perceived exertion for the walking task. Before incrementing the speed and continuing with the test, participants will be asked if participants would like to continue to walk and if the speed can be incremented. Participants metabolic and heart rate will be monitored frequently and recorded during this test. A physical exertion rating scale will be used to record participant's perceived exertion during every 2 minutes throughout the trial.
Change in Biomechanical Assessment [Gait Parameters and Surface Electromyography (EMG) Activation] Between Devices | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Surface EMG recording of specific muscles will be recorded during walking. The EMG electrodes detect electrical signals of the muscles. Reflective markers will be placed at specific locations on the upper and lower extremity joint/bony landmarks to record the motion while walking. The locations of the markers in space will be recorded by an infrared based multi-camera system during walking indoors on tile and over force plates.

SECONDARY OUTCOMES:
Change in Manual Muscle Test (MMT) | Week 1 (Pre-Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Muscle strength with be assessed using a hand held dynamometer for muscle strength testing of the lower limb
Change in Passive Range of Motion (PROM) | Week 1 (Pre-Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Lower extremity PROM and AROM will be measured using an electrogoniometer. This is a computerized device capable of measuring angles and giving an electronic output of the measurements. This device has been found to have high ratings of reliability and validity in the lower limb.
Change in Active Range of Motion (AROM) | Week 1 (Pre-Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Lower extremity AROM will be measured using an electrogoniometer. This is a computerized device capable of measuring angles and giving an electronic output of the measurements. This device has been found to have high ratings of reliability and validity in the lower limb.
6 Minute Walk Test (6MWT) with COSMED K4B2 Metabolic unit | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The 6 minute walk test is performed as an objective evaluation of functional exercise capacity. The test measures the distance that the patient can walk on a flat, hard surface, indoors, in a period of 6 minutes. The walk test is patient self-paced and assesses the level of functional capacity. Patients are allowed to stop and rest during the test, however, the timer does not stop. If the patient is unable to complete the time, the time stopped is noted and reason for stopping prematurely is recorded. This test will be administered while wearing a mask to measure oxygen consumption. COSMED K4B2 (K4B2 COSMED, Italy) is a portable gas analysis system that measures oxygen consumption (VO2) and Carbon-dioxide production (VCO2 ) in a breath by breath fashion.
Hill Assessment Index (HAI) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The Hill Assessment Index is a 12 point ordinal scale used to assess different gait patterns during ascent or descent of slopes. It was developed to detect differences in function with different knee units for transfemoral prosthetics. Time and oxygen consumption will be measured during ramp ascent and descent. These activities will be performed while wearing a mask to measure oxygen consumption. This test takes under 5 minutes to complete.
Stair Assessment Index (SAI) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The Stair Assessment Index is a 14 point ordinal scale originally used to assess functional abilities during ascent and descent of stairs. Time and oxygen consumption will be measured during stair ascent and descent. These activities will be performed while wearing a mask to measure oxygen consumption. These tests take under 5 minutes to complete.
Cross Walk Blinking Signal Test | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Time needed to cross a standard cross walk. The cross walk blinking signal test will measure how long it takes a participant to cross a designated street. The street that is designated for the test is 2 lanes and has ramps from the sidewalk to the street. The distance measured will be from the end of the ramp or edge of the curb on either side of the street. This distance is 36 feet. The literature recommends the cross walk velocity needed to safely cross is 0.9-1.2 m/s.
GAITRite® Data Capture | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The GAITRite® system automates measuring temporal and spatial gait parameters via an electronic walkway connected to a computer. The GAITRite® electronic walkway contains sensor pads encapsulated in a carpet to collect gait information. The system can be laid over any flat surface. The GAITRite® electronic walkway for the study shall be a minimum of 14 feet long. The GAITRite® data capture was chosen as measurement of the patient's overall gait quality. Patients will be asked to walk at a self-selected speed and fast speed across the GAITRite® electronic walkway.
5 Times Sit to Stand Test (5XSST) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The 5 Time Sit to Stand Test is a measure of functional lower limb strength during transitional movement. The individual sits in a standard height chair (43-45 cm) and is instructed to stand up and sit down 5 times as quickly as possible. The individual is not allowed to use upper extremities to push off and is instructed to cross arms over chest if able to do so. The test is scored by measuring the time it takes to complete the 5 stands. If the patient is unable to complete all 5 stands or requires assist greater than contact guard the test is scored as a fail.
4-Square Step Test | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Test of dynamic balance that clinically assesses the person's ability to step over objects forward, sideways and backwards. The test takes less than 5 minutes to administer and tests activity of daily living and motor skills.
Talks While Walking Test (TWWT- Dual task test) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The TWWT is used to determine the effects of cognitive attentional demands during walking by introducing a secondary thinking and talking task, while walking. Participants will perform the following tasks: timed walking up to 300 meters, performing a thinking and talking (numerical and/or vocabulary) task while sitting, and performing a thinking and talking task while walking (dual task) Participants voice will be recorded when performing all the thinking and talking tasks.
Outdoor Uneven Surfaces Test | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  This test will evaluate the participants gait characteristics and performance while walking on various surfaces that participants could encounter during activities of daily living. Participants will be asked to walk on typical outdoor uneven surfaces outside the entrance to the Rehabilitation Institute of Chicago (RIC), such as pavement, grass, uneven surfaces and ramps. Participants may use assistive device during this test. A researcher will walk with the participant to ensure safety and assist as needed.
Amputee Mobility Predictor | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  A tool used to predict the ambulatory potential of lower limb amputees, and measure function post-rehabilitation. It was developed to provide a more objective approach to rating amputees under the various K Classifications. The test can be performed with or without the prosthesis. The test involves activities of transfers, balance and walking. Score is out of 39 with each item scored in the range of 0-2
Mini Mental State Exam (MMSE) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  Is a brief screening tool to provide a quantitative assessment of cognitive impairment and to record cognitive changes over time. The MMSE consists of 11 simple questions or tasks grouped into 7 cognitive domains. A possible score of 30 is used to provide a picture of an individual's present cognitive performance based on direct observation of completion of test items/tasks.

OTHER OUTCOMES:
Modified Falls Efficacy Scale (mFES) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The mFES is self-report questionnaire consisting of 14 items which is designed to measure fear of falling in the elderly. It assesses an individual's perception of balance during activities of daily living by asking "how confident are you that you can do the following activities without falling."
Prosthesis Evaluation Questionnaire (PEQ) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The questionnaire was developed specifically to provide functional outcome measures in prosthetics that are more tuned to prosthesis-related changes in quality of life. It is a self-report questionnaire containing 54 questions organized into nine functional domain scales. Each of the scales may be used individually to measure only a specific domain of interest. The PEQ has been used in a wide variety of studies and is validated.
Orthotics & Prosthetics User Survey (OPUS) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The OPUS is a self-report questionnaire which is designed to evaluate the outcome of orthotic and prosthetic services. Three of the five domains will be administered: lower limb functional measure, health-related quality of life and satisfaction with device. The domains of upper limb functional measure and satisfaction with service are not applicable in this study.
World Health Organization Quality of Life (WHOQOL-BREF) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The WHOQOL-BREF is a self-report questionnaire that measures an individual's perceived quality of life. It contains four domains which cover physical health, psychological health, social relationships, and environment. Scores range from 0- 100 with 100 indicating a higher quality of life. The scores can be broken down by domain or taken as a whole. The WHOQOL-BREF is valid cross-culturally.
Numerical Pain Rating Scale (NPRS) | Week 1 (Pre-Assessment); Week 2 (Training Assessment); Week 3 (Training Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The NPRS is a measure of perceived pain intensity. It consists of asking a participant to assign a number to the pain experienced along a 0 (zero) to 10 (ten) scale, with 0 being "no pain" to 10 being "worst pain imaginable."
Socket Comfort Scale (SCS) | Week 1 (Pre-Assessment); Week 2 (Training Assessment); Week 3 (Training Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The Socket Comfort Scale quantifies the amputee's experience of pain and discomfort while wearing a prosthesis. It consists of asking the participant to assign a number to the pain/discomfort of participant along a 0 (zero) to 10 (ten) scale, with 0 represents the most uncomfortable socket fit you can imagine and 10 represents the most comfortable socket fit.
Prosthetic Limb Users Survey of Mobility™ (PLUS-M™) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The PLUS-M™ is a self-report instrument for measuring mobility of adults with lower limb amputation. It has been rigorously developed using modern psychometric methodology and is intended for use in clinical practice and research. PLUS-M™ instruments are based on a set of 44 calibrated questions called an item bank. PLUS-M™ instruments measure prosthetic users' mobility (i.e., the ability to move intentionally and independently from one place to another). PLUS-M™ questions assess respondents' perceived ability to carry out actions that require use of both lower limbs, ranging from household ambulation to outdoor recreational activities. The described activities relate to two primary forms of movement, locomotion (i.e., movement in a continuous, repeatable pattern) and/or postural transitions (i.e., movement from one position to another or one type of activity to another).
The Quebec User Evaluation of Satisfaction with Assistive Technology (QUEST) | Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  The QUEST is an instrument designed to measure the level of satisfaction attributed to assistive technologies. It does so using 27 variables which are scored in terms of perceived importance and satisfaction.
QUEBEC Back Pain Disability Scale | Week 1 (Pre-Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  This back pain scale is a self-reported measure that evaluates a patient's functional status related to back pain.
Borg Rate of Perceived Exertion (Borg RPE) | Week 1 (Pre-Assessment); Week 2 (Training Assessment); Week 3 (Training Assessment); Week 6-7 (Post-Training Assessments); Weeks 21-22 (Post-Training Assessment)
  A 6-20 item scale that measures perceived exertion during an activity.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Jayaraman, PT, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Shirley Ryan AbilityLab, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No